CLINICAL TRIAL: NCT04801849
Title: Vitamin E Dosing Study (VEDS): A Dose Finding Study of Vitamin E for the Treatment of Adult NAFLD
Brief Title: Vitamin E Dosing Study
Acronym: VEDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Duke University (Other); Liver Institute Northwest (Unknown); Indiana University (Other); St. Louis University (Other); University of California, San Diego (Other); University of Southern California (Other); University of California, San Francisco (Other); Virginia Commonwealth University (Other); The Cleveland Clinic (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10 VEDS; U24DK061730 (NIH); U01DK061732 (NIH); U01DK061713 (NIH); U01DK061737 (NIH); U01DK061728 (NIH); U01DK061718 (NIH); U01DK061734 (NIH); U01DK061738 (NIH); U01DK061731 (NIH); IRB00240822 (Other: JHM IRB)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
Keywords: Vitamin E; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double masked, placebo-controlled, parallel treatment groups
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vitamin E, 200 IU (Active Comparator): 200 IU of d-alpha tocopherol (vitamin E) taken once daily with breakfast
  Interventions: Drug: Vitamin E
- Vitamin E, 400 IU (Active Comparator): 400 IU of d-alpha tocopherol (vitamin E) taken once daily with breakfast
  Interventions: Drug: Vitamin E
- Vitamin E, 800 IU (Active Comparator): 800 IU of d-alpha tocopherol (vitamin E) taken once daily with breakfast
  Interventions: Drug: Vitamin E
- Placebo (Placebo Comparator): matching placebo taken once daily with breakfast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin E — Participants will be assigned to take 200 IU, 400 IU, or 800 IU of vitamin E in matching capsules daily for 24 weeks
  Other Names: d-alpha-tocopherol
  Arms: Vitamin E, 200 IU; Vitamin E, 400 IU; Vitamin E, 800 IU
Drug: Placebo — Participants will take a placebo vitamin E capsule daily for 24 weeks
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double masked, placebo-controlled, parallel treatment groups dosing trial of Vitamin E in adult nonalcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Adults age 18 years or older will be enrolled for 48 weeks and treated with 200 international units (IU), 400 IU, or 800 IU of Vitamin E or matching placebo for 24 weeks. The primary objective of the study is to determine the minimum effective dose of Vitamin E (d-alpha-tocopherol) based upon relative change in alanine aminotransferase (ALT) from baseline to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older as of the initial screening interview and provision of consent
* FibroScan CAP>280 dB/m within 60 days prior to randomization.
* ALT ≥ 60 U/L within 30 days of randomization

Exclusion Criteria:

* Concurrent or prior use (within 90 days) of vitamin E supplements in excess of 40 IU/day
* Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 g/day (~1.5 drinks/day) (> 10.5 drinks per week) in females and more than 30 g/day (~2 drinks/day) (>14 drinks per week) in males, respectively. One "standard" drink (or one alcoholic drink equivalent) contains roughly 14 grams of pure alcohol, which is found in: 12 ounces of regular beer, 5 ounces of wine, or 1.5 ounces of distilled spirits).
* Inability to reliably quantify alcohol consumption based upon local study physician judgment
* Continued use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins) for more than 2 weeks in the 6 months prior to randomization
* Current use of anticoagulation therapy (not including antiplatelet agents such as aspirin or clopidogrel)
* Platelet count below 150,000 /mm3 within 90 days of randomization
* History of condition(s) that cause increased risk of bleeding, including hemophilia A, hemophilia B, von Willebrand disease, or other clotting factor deficiencies.
* Prior or planned (during the study period) bariatric surgery (eg, gastroplasty, roux-en-Y gastric bypass)
* Uncontrolled diabetes defined as HbA1c 9.5% or higher within 60 days prior to randomization
* Clinical evidence of hepatic decompensation as defined by the presence of any of the following abnormalities:

  * Serum albumin less than 3.2 g/dL
  * International Normalized Ratio (INR) greater than 1.3
  * Direct bilirubin greater than 1.0 mg/dL
  * History of esophageal varices, ascites or hepatic encephalopathy
* Evidence of other forms of chronic liver disease:

  * Hepatitis B as defined by presence of hepatitis B surface antigen (HBsAg)
  * Hepatitis C as defined by presence of hepatitis C virus (HCV) RNA
  * Evidence of ongoing autoimmune liver disease as defined by compatible liver histology
  * Primary biliary cirrhosis as defined by the presence of at least 2 of these criteria (i) Biochemical evidence of cholestasis based mainly on alkaline phosphatase elevation (ii) Presence of anti-mitochondrial antibody (AMA) (iii) Histologic evidence of nonsuppurative destructive cholangitis and destruction of interlobular bile ducts[1]
  * Primary sclerosing cholangitis
  * Known history of Wilson disease, alpha-1-antitrypsin liver disease, or hemochromatosis. Any other type of liver disease that is currently active other than NASH such as drug-induced liver disease, liver cancer, or bile duct obstruction.
* Serum alanine aminotransferase (ALT) greater than 400 U/L within 90 days of randomization
* Moderate or severe renal impairment (serum creatinine ≥ 2.0 mg/dL or eGFR < 60 mg/mL/1.73m2)
* History of biliary diversion or evidence of current biliary obstruction
* Known positivity for Human Immunodeficiency Virus (HIV) infection
* Active, serious medical disease with likely life expectancy less than 5 years
* Active substance abuse including inhaled or injection drugs in the year prior to screening
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use ≥ 1 effective form(s) of birth control during the trial, breast feeding
* Current use of medications that may impact the absorption of fat-soluble vitamins (i.e. orlistat or cholestyramine)
* Pre-existing history of fat malabsorption
* Males at high risk of prostate cancer, including:

  * PSA >ULN at baseline
  * History of prostate cancer
  * Age 45 or older with a first-degree relative (father or brother) diagnosed with prostate cancer at an early age (younger than age 65).
  * Age 40 or older with more than one first-degree relative who had prostate cancer at an early age (younger than age 65)
* Participation in an IND trial in the 30 days before randomization
* Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study, including inability to swallow treatment capsules
* Failure or inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Relative change in alanine aminotransferase (ALT) from baseline to 24 weeks | 24 weeks
  ALT value in units/liter (U/L)

SECONDARY OUTCOMES:
Proportion of patients achieving normalization of alanine aminotransferase (ALT) at 24 weeks | 24 weeks
  Normalization of ALT (U/L) is defined as a decrease in ALT to less than or equal to the ULN at the 24 week visit among participants who had an ALT value greater than ULN at baseline. Values for upper limits of normal (ULN) are defined at each clinical center per institutional guidelines.
Mean change in serum alanine aminotransferase (ALT) from baseline | 24 weeks
  ALT value in U/L
Mean change in serum aspartate aminotransferase (AST) from baseline | 24 weeks
  AST value in U/L
Mean change in hepatic steatosis (fat in the liver) score determined by Fibroscan® Controlled Attenuation Parameter (CAP) software function | 24 weeks
  CAP (Control Attenuation Parameter) is expressed in decibels per meter (dB/m). This value is the median of all valid measurements performed during the examination. It ranges from 100 to 400 dB/m. Higher dB/m indicates worse liver fat.
  238 to 260 dB/m: 11% to 33% of liver with fatty change; 260 to 290 dB/m: 34% to 66% of liver with fatty change; 290 to 400 dB/m: at least 67% of liver with fatty change
Mean change in liver stiffness from baseline assessed by Fibroscan® | 24 weeks
  Fibroscan® measures stiffness in kiloPascal's (kPa) and ranges from 2 to 75. Normal range of FibroScan is between 2 to 7 kPa, and the average normal result is 5.3kPa. Higher kPa means more stiffness (scarring).

CONTACTS AND LOCATIONS:
Overall Officials: Arun Sanyal, MD, Principal Investigator — Virginia Commonwealth University
Locations (9):
- United States (9):
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University- Adults, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Virginia Commonwealth University, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the 2013 NIH Data Sharing Policy. Results and information from this trial will be submitted to ClinicalTrials.gov and a public use database deposited with the NIDDK Central Repository within two years of the date that the database is locked for analysis (interventional studies, primary and secondary outcomes).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data from this study may be requested from the NIDDK Central Repository (https://www.niddkrepository.org/search/study/) within two years of the date the database is locked for analysis (interventional studies, primary and secondary outcomes)
Access Criteria: Apply through the NIDDK Central Repository:
URL: https://repository.niddk.nih.gov/home

REFERENCES:
- See also: Nonalcoholic Steatohepatitis Clinical Research Network Centers — http://jhuccs1.us/nash/open/centers/centers.htm
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) — http://www2.niddk.nih.gov/